CLINICAL TRIAL: NCT04648995
Title: A Single-Blinded Split Face Prospective Study Comparing Different Energy, Efficacy, and Safety of UltraPulse CO2 Laser in the Treatment of Acne Scar Using Antera Quantitative 3D Image Analysis
Brief Title: TheTreatment of Acne Scar Using UltraPulse CO2 Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haute Beauté Skin & Vein Clinic (Other)
Collaborators: Lumenis Be Ltd. (Industry); Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Kuo-Liang Cheng, Superintendent, Haute Beauté Skin & Vein Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202007052
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-11

CONDITIONS: Acne Scar
Keywords: UltraPulse CO2 Laser; Antera Quantitative 3D Image; Collagen; Elastic fiber; Scale for global severity of facial acne scar

STUDY DESIGN:
Intervention Model Description: Low energy:
  Half of the face that receives low energy, their central base of boxcar scar will be treated with 20mJ, while shoulder of scar will be treated with 50 mJ
  High energy:
  Half of the face that receives low energy, their central base of boxcar scar will be treated with 30mJ, while shoulder of scar will be treated with 60 mJ
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High energy (Other): Half of the face that receives low energy, their central base of boxcar scar will be treated with 30mJ, while shoulder of scar will be treated with 60 mJ
  Interventions: Device: High energy (UltraPulse)
- Low energy (Other): Half of the face that receives low energy, their central base of boxcar scar will be treated with 20mJ, while shoulder of scar will be treated with 50 mJ
  Interventions: Device: Low energy (UltraPulse)

INTERVENTIONS:
Device: High energy (UltraPulse) — Half of the face that receives low energy, their central base of boxcar scar will be treated with 30mJ, while shoulder of scar will be treated with 60 mJ
  Arms: High energy
Device: Low energy (UltraPulse) — Half of the face that receives low energy, their central base of boxcar scar will be treated with 20mJ, while shoulder of scar will be treated with 50 mJ
  Arms: Low energy

SUMMARY:
Purpose of the study is to assess the effect and evaluate topographic volume changes of UltraPulse at treating boxcar scars with different energy and the effect of UltraPulse at treating icepick scars.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 24 hour screening period to determine eligibility for study entry. Upon enrollment, patient who fulfill all the inclusion criteria and does not fulfill any exclusion criteria will be scheduled for their visits.

All subjects will be receiving two sessions of treatment, with the two sessions 8-12 weeks apart. Subjects' face will be divided to left and right, with each side randomized to receive a low versus high energy setting. In the low energy setting side of the face, central base of boxcar scar will be treated with 20mJ, while shoulder of scar will be treated with 50 mJ. In the high energy setting side of the face, central base of boxcar scar will be treated with 30mJ, while shoulder of scar will be treated with 60 mJ. Subject will be blinded regarding which side of the face received low versus high energy setting.

Ultrasound will be used to assess epidermal and dermal thickness change at the treated area. This will be performed before the 1st and 2nd treatment session as well as one month and three month after the 2nd treatment session.

Antera Quantitative 3D Image Analysis will be performed before and after the 1st and 2nd treatment session as well as one month and three month after the 2nd treatment session.

3mm punch biopsy will be taken from 10 volunteers over bilateral face before the 1st treatment session and 3 month after the 2nd treatment session (total of 4 sample will be obtained in each volunteer). Skin specimen will be stained with hematoxylin and eosin as well as relevant stain for collagen and elastic fiber.

Clinical photograph will be taken before and after the 1st and 2nd treatment session as well as one month and three month after the 2nd treatment session. Two blinded board certified dermatologist will be asked to rate the improvement of acne scar by GSAAS according to the clinical photograph taken.

All subjects will be asked to rate their satisfaction regarding treatment response over each side of the face using a 0 to 10 point scale chart.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have to be aged from 20 to 60 year-old
* Subjects currently have an area of involvement approximately 2cm × 2cm on each side of the face over the temples or cheek bone area
* Classified as mild to moderate acne scar according to global severity of facial acne scar (GSAAS) score
* After evaluation by clinician, those subjects to be treated with "Lumenis"CO2 Laser System (UltraPulse) can benefit from this laser treatment
* Subjects need to be fully functional and aware of the pros and cons of the study. Subject is capable to make self judgement and sign the inform consent under his/her own will
* Others: Have fully understand about this study and is willing to cooperate with the instruction of the study

Exclusion Criteria:

* Those who were known to have keloid formation
* Those who have porphyria or known photosensitivity
* Those who previously underwent laser therapy treatment or skin biopsy and have showed poor result or adverse effect
* Those who were classified as "severe" according to GSAAS system
* Those who have bleeding tendency
* Those who present with clinical data suggesting abnormal platelet function or coagulation disorder (such as prolonged aPTT or PT)
* Those that are currently taking anticoagulants or anti-platelet drugs
* Those who are on aspirin or other NSAIDs
* Those who have history of granulomatous or connective tissue disease
* Female subjects with a positive pregnancy test
* Women who refuse to stay on effective contraception or refuse pregnancy tests during the study
* After evaluation by the clinician, those that have been enrolled in clinical studies over the past 6 months that may alter the current study result
* After evaluation by the clinician, those currently or had previous treatment of atrophic acne scars with fillers, lasers, deep chemical peels, or any other medical or surgical treatment which in the investigators' opinion could alter the results of the current clinical study
* Those that are currently taking photo-sensitive drugs, oral isotretinoin, iron supplement or other herbal medication
* Those that have received laser treatment over the lesion area over the past 3 months
* Those that are currently pregnant or breastfeeding
* After evaluation by the clinician, and concluded underline epilepsy, area to be treated is under infection or ulceration, poor wound healing)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-09-08 (Estimated); Study Completion 2021-11-28 (Estimated)

PRIMARY OUTCOMES:
Topographic volume changes of acne scars from baseline one month and three month after the 2nd treatment session | from baseline one month and three month after the 2nd treatment session
  Topographic volume changes of acne scars from baseline one month and three month after the 2nd treatment session
Histological change in epidermal/dermal component including elastic fiber and collagen synthesis three month after the 2nd treatment session from baseline | three month after the 2nd treatment session from baseline
  Histological change in epidermal/dermal component including elastic fiber and collagen synthesis three month after the 2nd treatment session from baseline

SECONDARY OUTCOMES:
Access improvement of acne scar by Scale for global severity of facial acne scar from baseline one month and three month after the 2nd treatment session in both the low and high energy treated arm | from baseline one month and three month after the 2nd treatment session
  Access improvement of acne scar by Scale for global severity of facial acne scar from baseline one month and three month after the 2nd treatment session in both the low and high energy treated arm. The minimum and maximum values of Scale for global severity of facial acne scar are 0 and 5, and higher scores mean a worse outcome.
Compare the difference of improvement of acne scar by Scale for global severity of facial acne scar in the low versus high energy treated arm | from baseline and three month after the 2nd treatment session
  Compare the difference of improvement of acne scar by Scale for global severity of facial acne scar in the low versus high energy treated arm. The minimum and maximum values of Scale for global severity of facial acne scar are 0 and 5, and higher scores mean a worse outcome.
Compare the difference of newly synthesis collagen and elastic fiber through staining in the low versus high energy treated arm | from baseline and three month after the 2nd treatment session
  Compare the difference of newly synthesis collagen and elastic fiber through staining in the low versus high energy treated arm
Assess the frequency and severity of encountered side effects in the low versus high energy treated arm | from baseline and three month after the 2nd treatment session
  Assess the frequency and severity of encountered side effects in the low versus high energy treated arm
Subjects' satisfaction score rated in a 0 to 10 point scale | after the 2nd treatment session、one month and three month after the 2nd treatment session
  Subjects' satisfaction score rated in a 0 to 10 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Liang Cheng, MD, Principal Investigator — Haute Beauté Skin & Vein Clinic
Locations (1):
- HAUTE BEAUTÉ Skin & Vein Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dreno B, Thiboutot D, Layton AM, Berson D, Perez M, Kang S; Global Alliance to Improve Outcomes in Acne. Large-scale international study enhances understanding of an emerging acne population: adult females. J Eur Acad Dermatol Venereol. 2015 Jun;29(6):1096-106. doi: 10.1111/jdv.12757. Epub 2014 Oct 8. PMID 25296739
- [Background] Bhargava S, Kumar U, Varma K. Subcision and Microneedling as an Inexpensive and Safe Combination to Treat Atrophic Acne Scars in Dark Skin: A Prospective Study of 45 Patients at a Tertiary Care Center. J Clin Aesthet Dermatol. 2019 Aug;12(8):18-22. Epub 2019 Aug 1. PMID 31531167
- [Background] Jacob CI, Dover JS, Kaminer MS. Acne scarring: a classification system and review of treatment options. J Am Acad Dermatol. 2001 Jul;45(1):109-17. doi: 10.1067/mjd.2001.113451. PMID 11423843
- [Background] Alster TS, Li MKY. Microneedling of Scars: A Large Prospective Study with Long-Term Follow-Up. Plast Reconstr Surg. 2020 Feb;145(2):358-364. doi: 10.1097/PRS.0000000000006462. PMID 31985622
- [Background] Arsiwala SZ, Desai SR. Fractional Carbon Dioxide Laser: Optimizing Treatment Outcomes for Pigmented Atrophic Acne Scars in Skin of Color. J Cutan Aesthet Surg. 2019 Apr-Jun;12(2):85-94. doi: 10.4103/JCAS.JCAS_171_18. PMID 31413476
- [Background] Emer J. Platelet-Rich Plasma (PRP): Current Applications in Dermatology. Skin Therapy Lett. 2019 Sep;24(5):1-6. PMID 31584784
- [Background] Mu YZ, Jiang L, Yang H. The efficacy of fractional ablative carbon dioxide laser combined with other therapies in acne scars. Dermatol Ther. 2019 Nov;32(6):e13084. doi: 10.1111/dth.13084. Epub 2019 Oct 7. PMID 31496020
- [Background] Tanizaki H, Tanioka M, Yamashita Y, Hayashi N. Quantitative evaluation of atrophic acne scars using 3D image analysis with reflected LED light. Skin Res Technol. 2020 Jan;26(1):20-24. doi: 10.1111/srt.12756. Epub 2019 Sep 2. PMID 31478266
- [Background] Petit L, Zugaj D, Bettoli V, Dreno B, Kang S, Tan J, Torres V, Layton AM, Martel P. Validation of 3D skin imaging for objective repeatable quantification of severity of atrophic acne scarring. Skin Res Technol. 2018 Nov;24(4):542-550. doi: 10.1111/srt.12464. Epub 2018 Mar 6. PMID 29512189